CLINICAL TRIAL: NCT01096784
Title: Determination of the rhIGF-1/rhIGFBP-3 Dose, Administered as a Continuous Infusion, Required to Establish and Maintain Longitudinal Serum IGF-1 Levels Within Physiological Levels in Premature Infants, to Prevent Retinopathy of Prematurity A Phase 2, Randomized Controlled, Assessor-blind, Dose Confirming, Pharmacokinetic, Safety and Efficacy, Multicenter Study
Brief Title: IGF-1/IGFBP3 Prevention of Retinopathy of Prematurity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ROPP-2008-01; 2007-007872-40 (EudraCT Number)
Record Dates: First submitted 2010-03-09; First posted 2010-03-31 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Retinopathy of Prematurity (ROP)
Keywords: insulin-like growth factor; ROP; IGF-I; BPD; bronchopulmonary dysplasia; retinopathy of prematurity
MeSH Terms: conditions — Retinopathy of Prematurity; Bronchopulmonary Dysplasia | interventions — Insulin-Like Growth Factor I

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhIGF-I/rhIGFBP-3 (Active Comparator): Continuous IV Infusion
  Interventions: Drug: rhIGF-I/rhIGFBP-3
- Control (No Intervention): The comparator group will receive no treatment with rhIGF-1/rhIGFBP-3

INTERVENTIONS:
Drug: rhIGF-I/rhIGFBP-3 — Continuous intravenous infusion
  Other Names: Mecasermin Rinfabate
  Arms: rhIGF-I/rhIGFBP-3

SUMMARY:
To compare the severity of retinopathy of prematurity (ROP) among treated infants with an untreated control population, matched for gestational age at birth while confirming the dose of rhIGF-1/rhIGFBP-3 is safe and efficacious.

DETAILED DESCRIPTION:
When preterm infants are deprived of their natural intrauterine environment they lose access to important factors, normally found in utero, such as proteins, growth factors, and cytokines. It has been demonstrated that insulin-like growth factor-1 (IGF-1) is one such factor. In utero these biological factors are introduced to the fetus via placental absorption or ingestion from amniotic fluid. Deprivation of such factors is likely to cause inhibition or improper stimulation of important pathways, which in the case of the eye may cause abnormal retinal vascular growth, the hallmark of retinopathy of prematurity (ROP).

Retinopathy of prematurity is the major cause of blindness in children in the developed and developing world, despite the availability of current treatment of late-stage ROP. As developing countries provide more neonatal and maternal intensive care, which increases the survival of preterm born infants, the incidence of ROP is increasing.

This phase 2 study was originally designed in 3 sections, Sections A, B, and C which are now complete. The protocol was amended and patients enrolled from this point forward will be enrolled into Section D.

In Study Section D, a total of 120 subjects (GA of 23 weeks + 0 days to 27 weeks + 6 days) will be randomly assigned with 1:1 allocation ratio to either treatment with rhIGF-1/rhIGFBP-3 or to receive standard neonatal care (Control Group) to obtain at least 80 evaluable subjects. Duration of infusion will last at longest from Study Day 0 (day of birth) up to and including PMA 29 weeks + 6 days, when the subject's endogenous production of IGF-1 is considered sufficient to maintain physiologic serum IGF-1 levels. After discontinuation of study drug infusion, each subject will be followed to PMA 40 weeks ± 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parents/guardians;
* Subject must be between GA of 26 weeks + 0 days and 27 weeks + 6 days (Study Section A) or between GA of 23 weeks + 0 days and 27 weeks + 6 days (Study Sections B, C, and D), inclusive

Exclusion Criteria:

* Subjects born small for gestational age (SGA), ie, body weight at birth <-2 standard deviation score (SDS) (Study Section A only)
* Detectable gross malformation
* Known or suspected chromosomal abnormality, genetic disorder, or syndrome, according to the Investigator's opinion
* Persistent blood glucose level <2.5 mmol/L or >10 mmol/L at Study Day 0 (day of birth) to exclude severe congenital abnormalities of glucose metabolism
* Anticipated need of administration of erythropoietin (rhEPO) during treatment with study drug.
* Any maternal diabetes requiring insulin during the pregnancy
* Clinically significant neurological disease according to the Investigator's opinion(Stage 1 IVH allowed)
* Any other condition or therapy that, in the Investigator's opinion, may pose a risk to the subject or interfere with the subject's ability to be compliant with this protocol or interfere with interpretation of results
* Monozygotic twins
* Subject participating or plans to participate in a clinical study of another investigational study drug

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2010-06-18 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (24):
- United States (8):
  - University of South Alabama Children's and Women's Hospital, Mobile, Alabama
  - Univ of California Irvine Med Center, Irvine, California
  - Georgia Regents Medical Center, Augusta, Georgia
  - Univ of Mississippi Medical Center, Jackson, Mississippi
  - Vidant Medical Center, Greenville, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
- Italy (4):
  - D.A.I. Materno Infantile, S.O.D. Neonatologia e Terapia Intensiva Neonatale - Azienda Ospedaliero-Universitaria Careggi, Florence
  - U.O.C Patologia e Terapia Intensiva Neonatale, Istituto Giannina Gaslini-Istituto Pediatrico di Ricovero e Cura a Carattere Scientifico, Genova
  - University of Padua, Padua
  - Dipartimento per la Tutella della Salute della Donna e della Vita Nascente, del Bambino e dell'Adolescente-U.O.C. Neonatologia-Poli. Gemelli, Rome
- VU medical Center, Amsterdam, Netherlands
- Poland (2):
  - Instytut Centrum Zdrowia Matki Polki, Lódz
  - Ginekologiczno-Położniczy Szpital Kliniczny Uniwersytetu Medycznego w Poznani, Poznan
- Sweden (2):
  - Skånes University Hospital Lund, Lund
  - Karolinska Universtitetssjukhuset i Huddinge, Stockholm
- United Kingdom (7):
  - Addenbrookes Hospital, Cambridge
  - St Peter's Hospital; Ashford & S, Chertsey
  - University Hospital, Coventry
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - UCL EGA Institute for Women's Health, London
  - St. Mary's Hospital, Manchester
  - Norfolk and Norwich University, Norwich

REFERENCES:
- [Background] Lofqvist C, Niklasson A, Engstrom E, Friberg LE, Camacho-Hubner C, Ley D, Borg J, Smith LE, Hellstrom A. A pharmacokinetic and dosing study of intravenous insulin-like growth factor-I and IGF-binding protein-3 complex to preterm infants. Pediatr Res. 2009 May;65(5):574-9. doi: 10.1203/PDR.0b013e31819d9e8c. PMID 19190540
- [Result] Ley D, Hansen-Pupp I, Niklasson A, Domellof M, Friberg LE, Borg J, Lofqvist C, Hellgren G, Smith LE, Hard AL, Hellstrom A. Longitudinal infusion of a complex of insulin-like growth factor-I and IGF-binding protein-3 in five preterm infants: pharmacokinetics and short-term safety. Pediatr Res. 2013 Jan;73(1):68-74. doi: 10.1038/pr.2012.146. Epub 2012 Oct 24. PMID 23095978
- [Derived] Klevebro S, Hellgren G, Hansen-Pupp I, Wackernagel D, Hallberg B, Borg J, Pivodic A, Smith L, Ley D, Hellstrom A. Elevated levels of IL-6 and IGFBP-1 predict low serum IGF-1 levels during continuous infusion of rhIGF-1/rhIGFBP-3 in extremely preterm infants. Growth Horm IGF Res. 2020 Feb;50:1-8. doi: 10.1016/j.ghir.2019.11.001. Epub 2019 Nov 9. PMID 31756675
- [Derived] Ley D, Hallberg B, Hansen-Pupp I, Dani C, Ramenghi LA, Marlow N, Beardsall K, Bhatti F, Dunger D, Higginson JD, Mahaveer A, Mezu-Ndubuisi OJ, Reynolds P, Giannantonio C, van Weissenbruch M, Barton N, Tocoian A, Hamdani M, Jochim E, Mangili A, Chung JK, Turner MA, Smith LEH, Hellstrom A; study team. rhIGF-1/rhIGFBP-3 in Preterm Infants: A Phase 2 Randomized Controlled Trial. J Pediatr. 2019 Mar;206:56-65.e8. doi: 10.1016/j.jpeds.2018.10.033. Epub 2018 Nov 22. PMID 30471715
- [Derived] Hansen-Pupp I, Hellstrom A, Hamdani M, Tocoian A, Kreher NC, Ley D, Hallberg B. Continuous longitudinal infusion of rhIGF-1/rhIGFBP-3 in extremely preterm infants: Evaluation of feasibility in a phase II study. Growth Horm IGF Res. 2017 Oct;36:44-51. doi: 10.1016/j.ghir.2017.08.004. Epub 2017 Aug 31. PMID 28934640
- [Derived] Chung JK, Hallberg B, Hansen-Pupp I, Graham MA, Fetterly G, Sharma J, Tocoian A, Kreher NC, Barton N, Hellstrom A, Ley D. Development and verification of a pharmacokinetic model to optimize physiologic replacement of rhIGF-1/rhIGFBP-3 in preterm infants. Pediatr Res. 2017 Mar;81(3):504-510. doi: 10.1038/pr.2016.255. Epub 2016 Nov 21. PMID 27870826
- [Derived] Lundgren P, Stoltz Sjostrom E, Domellof M, Kallen K, Holmstrom G, Hard AL, Smith LE, Lofqvist C, Hellstrom A. WINROP identifies severe retinopathy of prematurity at an early stage in a nation-based cohort of extremely preterm infants. PLoS One. 2013 Sep 12;8(9):e73256. doi: 10.1371/journal.pone.0073256. eCollection 2013. PMID 24069180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in multiple centres in Italy, the Netherlands, Poland, Sweden, the United Kingdom and the United States between 18 Jun 2010 and 30 March 2016.
Pre-assignment Details: A total of 121 participants were enrolled and randomized into the study.
Groups:
- rhIGF-1/rhIGFBP-3: Participants received insulin-like growth factor (rhIGF-I)/insulin-like growth factor binding protein-3 (rhIGFBP-3) 250 microgram per kilogram (mcg/kg) for 24 hours through continuous intravenous (IV) infusion from Day 0 up to 29 weeks 6 days of post-menstrual age (PMA).
- Standard of Care (Control): Participants in this control group do not received any treatment other than the standard care.
Period: Overall Study
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Started | 61 | 60
Completed | 46 | 46
Not Completed | 15 | 14
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 11 | 9
Not completed — Protocol Deviation | 2 | 2
Not completed — Administrative Decision | 0 | 1
Not completed — Other Unspecified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) set included all enrolled participants for whom a randomization number was assigned.
Groups:
- rhIGF-1/rhIGFBP-3: Participants received rhIGF-I/rhIGFBP-3 250 mcg/kg for 24 hours through continuous IV infusion from Day 0 up to 29 weeks 6 days of PMA.
- Total: Total of all reporting groups
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control) | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 25.60 (1.207) | 25.62 (1.397) | 25.61 (1.300)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Severity of Retinopathy of Prematurity (ROP) as Compared to the Severity of ROP in an Untreated Control Population
Description: ROP was measured by central exams with fundus photography. Maximum severity of ROP stage across all retinal examinations included International Classification of Retinopathy of Prematurity, a 5 stage system, for the classification of ROP with 7 different outcomes of the ROP stage in each retinal examination: 0, 1, 2, 3, 3+, 4, and 5. This is an ordinal scale with higher numbers indicating a more severe outcome. The maximum severity of ROP across all time points was assessed from 31 PMA weeks up to 40 PMA Weeks +/- 4 days (end of study).
Time Frame: End of study
Population: Full Analysis Set (FAS) included all randomized participants who received the study drug and participants in the control group who received Standard of Care.
Measure: Number; unit: participants
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
participants
  ROP of Stage "0" | 14 | 24
  ROP of Stage "1" | 4 | 4
  ROP of Stage "2" | 17 | 13
  ROP of Stage "3" | 6 | 3
  ROP of Stage "3+" | 6 | 6
  ROP of Stage "4" | 0 | 0
  ROP of Stage "5" | 0 | 0
  Missing | 14 | 10
Statistical Analysis 1: Comparison: rhIGF-1/rhIGFBP-3 vs Standard of Care (Control); Test type: Superiority or Other; p = 0.0642, CMH Row Mean Score Test

2. Secondary Outcome: Time to Discharge From Neonatal Intensive Care (TDNIC)
Time Frame: Day 0 to 40 Weeks Post Menstrual Age (EOS)
Population: FAS with number of participants evaluable for this outcome.
Measure: Median (Full Range); unit: Days
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 37 | 31
Days | 82.00 [69.00 to 96.00] | 74.00 [69.00 to 93.00]

3. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD)
Description: Severity of BPD as mild, moderate and severe were based on the National Institute of Child Health and Human Development (NICHD) guidelines for preterm infants born at gestational age (GA) less than (<) 32 weeks. Mild: oxygen requirement during the first 28 days but in room air at PMA 36 weeks or discharge to home, whichever comes first. Moderate BPD: oxygen requirement during the first 28 days and oxygen <30 percent (%) at PMA 36 weeks or discharge to home, whichever comes first. Severe BPD: oxygen requirement during the first 28 days and oxygen greater than equal (≥)30% through head hood or nasal canula, or continuous positive airway pressure, or mechanical ventilation, or high flow nasal cannula ≥2 L/min at PMA 36 weeks or discharge to home, whichever comes first.
Time Frame: At 36 Weeks Post Menstrual Age
Population: FAS with participants evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 47 | 49
participants
  No BPD | 4 | 4
  Mild | 23 | 16
  Moderate | 9 | 5
  Severe | 10 | 22
  Unable to determine | 1 | 2

4. Secondary Outcome: Rate of Change in Body Weight
Description: The rate of change is the rate of specific body weight change per day in kilogram (kg).
Time Frame: Day 0 to 40 Weeks Post Menstrual Age (EOS)
Population: FAS
Measure: Mean (95% Confidence Interval); unit: kilogram per day (kg/day)
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
kilogram per day (kg/day) | 0.021 [0.019 to 0.022] | 0.023 [0.021 to 0.024]

5. Secondary Outcome: Rate of Change in Length
Description: The rate of change is the length change per day in centimeter (cm).
Time Frame: Day 0 to 40 Weeks Post Menstrual Age (EOS)
Population: FAS
Measure: Mean (95% Confidence Interval); unit: centimeter per day (cm/day)
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
centimeter per day (cm/day) | 0.141 [0.0132 to 0.149] | 0.156 [0.147 to 0.164]

6. Secondary Outcome: Rate of Change in Head Circumference
Description: The rate of change is the head circumference change per day in centimetre (cm).
Time Frame: Day 0 to 40 Weeks Post Menstrual Age (EOS)
Population: FAS
Measure: Mean (95% Confidence Interval); unit: cm/day
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
cm/day | 0.115 [0.109 to 0.121] | 0.119 [0.113 to 0.125]

7. Secondary Outcome: Brain Development Assessed by Brain Volume at 40 Weeks PMA/EOS
Description: Brain volume was measured using cerebral magnetic resonance imaging (MRI). Brain volume included cerebrospinal volume, gray matter volume, white matter volume, and total cerebellar volume
Time Frame: 40 Weeks PMA/ (EOS) +/- 4 days
Population: FAS
Measure: Mean (Standard Deviation); unit: cubic centimeter
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
cubic centimeter
  Cerebrospinal Fluid Volume: number analyzed (Participants) | 45 | 40
  Cerebrospinal Fluid Volume | 87.94 (26.788) | 93.70 (25.540)
  Gray Matter Volume: number analyzed (Participants) | 45 | 40
  Gray Matter Volume | 206.34 (31.797) | 221.98 (33.827)
  White Matter Volume: number analyzed (Participants) | 45 | 40
  White Matter Volume | 110.23 (25.565) | 117.62 (24.422)
  Total Cerebellar Volume: number analyzed (Participants) | 45 | 41
  Total Cerebellar Volume | 18.27 (5.302) | 19.20 (4.854)

8. Secondary Outcome: Percentage of Participants With Intraventricular Hemorrhage (IVH)
Description: Development of intraventricular hemorrhage was assessed by cerebral ultrasound and coded as a binary endpoint (presence or absence of IVH).
Time Frame: Day 0 to 40 Weeks Post Menstrual Age (EOS)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
percentage of participants
  Yes | 19.67 | 30.0
  No | 80.33 | 70.0

9. Secondary Outcome: Area Under Curve for Maximum Severity of ROP Stage (AUC for ROP)
Description: Integration of the maximum severity of ROP stage and the duration of the time interval with respect to each retinal examination. AUC for the maximum severity of ROP was calculated using the trapezoidal rule. The area between each 2 visits was calculated by multiplying the average of the maximum severities of the 2 visits by the difference in days and analyzed using the van Elteren test. ROP is classified according to the International Classification and is subdivided into 5 stages (1-5) with higher values representing greater severity.
Time Frame: Every 1-2 weeks starting at 31 weeks PMA/ EOS +/- 4 days
Population: Full analysis set with number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: ROP severity score*days
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 42 | 49
ROP severity score*days | 47.95 (47.384) | 32.17 (40.151)

10. Secondary Outcome: Percentage of Participants With Maximum Severity of ROP Stage Greater Than or Equal to 3 at Any Time During the Study
Description: ROP was measured by central exams with fundus photography. Maximum severity of ROP stage across all retinal examinations included International Classification of Retinopathy of Prematurity, a 5 stage system, for the classification of ROP with 7 different outcomes of the ROP stage in each retinal examination: 0, 1, 2, 3, 3+, 4, and 5. This is an ordinal scale with higher numbers indicating a more severe outcome.
Time Frame: Day 0 to 40 Weeks Post Menstrual Age (EOS)
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
Percentage of participants
  Yes | 25.53 | 18.00
  No | 74.47 | 82.00

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAE) and Treatment Emergent Serious Adverse Event (TESAE)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse event was defined as the onset of any AE or if the severity of a pre-existing AE worsened any time on or after the date of first dose of investigational product.
Time Frame: Day 0 to 40 Weeks Post Menstrual Age (EOS)
Population: Safety Analysis Set (SAF) included all randomized participants who received the study drug and participants in the control group who received standard of care, and for whom at least 1 safety assessment was completed.
Measure: Number; unit: participants
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
participants
  Participants with TEAE | 60 | 60
  Participants with TESAE | 48 | 37

12. Secondary Outcome: Percentage of Serum IGF-1 Concentrations Falling Within Target Range After Infusion of rhIGF-1/rhIGFBP-3
Description: Serum samples were collected from treated and control participants for quantification of IGF-1 using validated immunoassays. Target range of serum IGF-1 was 28-109 mcg/L. The percentage of serum IGF-1 levels across treated participants that fall within the range was reported.
Time Frame: Day 0 to 40 Weeks Post Menstrual Age (EOS)
Population: FAS was analysed.
Measure: Number; unit: percentage of serum concentration
Groups:
- rhIGF-I/rhIGFBP-3: Participants received rhIGF-I/rhIGFBP-3 250 mcg/kg for 24 hours through continuous IV infusion from Day 0 up to 29 weeks 6 days of PMA.
- Control: Participants in this control group do not received any treatment other than the standard care.
Arm/Group | rhIGF-I/rhIGFBP-3 | Control
Number analyzed (Participants) | 61 | 60
percentage of serum concentration | 66.23 | 6.28

13. Secondary Outcome: Serum Concentrations of IGFBP-3 After Intravenous (IV) Infusion of rhIGF-1/rhIGFBP-3
Time Frame: Day 0 and Week 40 Post Menstrual Age
Population: FAS.
Measure: Mean (Standard Deviation); unit: microgram per liter
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
microgram per liter
  Day 0: number analyzed (Participants) | 60 | 60
  Day 0 | 494.2 (200.38) | 469.9 (180.52)
  Week 40: number analyzed (Participants) | 47 | 46
  Week 40 | 830.1 (200.17) | 882.1 (274.43)

14. Secondary Outcome: Serum Concentrations of Acid Labile Sub-unit (ALS) After Intravenous (IV) Infusion of rhIGF-1/rhIGFBP-3
Time Frame: Day 7 and Week 40 Post Menstrual Age
Population: FAS.
Measure: Mean (Standard Deviation); unit: microgram per liter
Arm/Group | rhIGF-1/rhIGFBP-3 | Standard of Care (Control)
Number analyzed (Participants) | 61 | 60
microgram per liter
  Day 7: number analyzed (Participants) | 60 | 60
  Day 7 | 411.9 (237.91) | 500.3 (350.59)
  Week 40: number analyzed (Participants) | 47 | 46
  Week 40 | 1804.6 (629.61) | 2114.3 (941.94)

ADVERSE EVENTS:
Time Frame: From Day 0 upto 4 days from PMA 40 Weeks
Arm/Group | rhIGF-I/rhIGFBP-3 | Standard of Care (Control)
Serious Adverse Events (participants affected / at risk) | 48/61 | 37/60
Other Adverse Events (participants affected / at risk) | 58/61 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhIGF-I/rhIGFBP-3 (N=61) | Standard of Care (Control) (N=60)
Coagulation disorder neonatal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neonatal hypotension (Vascular disorders) | 2 (2) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 5 (6) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Intra-Abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Meconium ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 6 (6) | 3 (3)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 13 (13) | 14 (14)
Bradycardia neonatal (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Citrobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 3 (3)
Group b streptococcus neonatal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Neonatal pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 7 (8) | 1 (1)
Serratia sepsis (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 9 (10) | 7 (9)
Pco2 increased (Investigations) | 0 (0) | 1 (1)
Renal failure neonatal (Renal and urinary disorders) | 3 (3) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage neonatal (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion neonatal (Nervous system disorders) | 2 (2) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 7 (8) | 8 (8)
Periventricular leukomalacia (Nervous system disorders) | 4 (4) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (8)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 9 (13)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhIGF-I/rhIGFBP-3 (N=61) | Standard of Care (Control) (N=60)
Anaemia neonatal (Blood and lymphatic system disorders) | 46 (210) | 44 (157)
Coagulation disorder neonatal (Blood and lymphatic system disorders) | 9 (10) | 8 (12)
Neutropenia neonatal (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 12 (15) | 9 (13)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Osteopenia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9)
Neonatal hypotension (Vascular disorders) | 23 (33) | 15 (27)
Retinopathy of prematurity (Eye disorders) | 39 (106) | 37 (89)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (9) | 6 (6)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 3 (3)
Inguinal hernia (Gastrointestinal disorders) | 9 (10) | 11 (11)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 6 (6)
Vomiting neonatal (Gastrointestinal disorders) | 2 (2) | 3 (5)
Generalised oedema (General disorders) | 9 (15) | 4 (5)
Infusion site extravasation (General disorders) | 1 (1) | 3 (8)
Oedema peripheral (General disorders) | 9 (11) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 6 (6) | 9 (10)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 53 (67) | 45 (57)
Bradycardia neonatal (Cardiac disorders) | 13 (18) | 5 (6)
Neonatal tachycardia (Cardiac disorders) | 4 (8) | 0 (0)
Fungal skin infection (Infections and infestations) | 3 (6) | 3 (6)
Neonatal pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 4 (4) | 5 (6)
Rhinitis (Infections and infestations) | 4 (5) | 3 (6)
Sepsis neonatal (Infections and infestations) | 16 (33) | 15 (29)
Staphylococcal sepsis (Infections and infestations) | 9 (14) | 12 (16)
Blood alkaline phosphatase increased (Investigations) | 5 (6) | 6 (6)
C-Reactive protein increased (Investigations) | 5 (6) | 4 (5)
Oliguria (Renal and urinary disorders) | 5 (5) | 3 (4)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 12 (14) | 14 (18)
Neonatal cholestasis (Hepatobiliary disorders) | 2 (2) | 6 (6)
Acidosis (Metabolism and nutrition disorders) | 4 (5) | 8 (9)
Feeding disorder neonatal (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 24 (41) | 28 (55)
Hypernatraemia (Metabolism and nutrition disorders) | 6 (7) | 11 (13)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (6) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (20) | 6 (6)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 18 (22) | 19 (27)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (24) | 11 (18)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Metabolic acidosis (Metabolism and nutrition disorders) | 17 (43) | 22 (46)
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 23 (43) | 22 (39)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 3 (3)
Convulsion neonatal (Nervous system disorders) | 3 (3) | 3 (3)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 11 (13) | 18 (19)
Periventricular leukomalacia (Nervous system disorders) | 1 (1) | 3 (3)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 28 (34) | 30 (38)
Poor weight gain neonatal (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4)
Oedema genital (Reproductive system and breast disorders) | 8 (9) | 1 (2)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 34 (37) | 37 (42)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (11)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (5)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 26 (42) | 16 (32)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 13 (21)
Neonatal respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 10 (30) | 5 (11)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 27 (31) | 32 (41)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 5 (5)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (11)
Pulmonary oedema neonatal (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.